CLINICAL TRIAL: NCT01073007
Title: Multicentric, Randomized, Double-blind Clinical Trial to Evaluate the Efficacy of Simvastatin in the Acute Phase of Ischemic Stroke
Brief Title: Stroke Treatment With Acute Reperfusion and Simvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STARS07; EC07/90195 (Other: Fondo de Investigación Sanitaria)
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2014-06

CONDITIONS: Stroke, Acute
Keywords: Acute Stroke; tissue plasminogen activator; simvastatin
MeSH Terms: conditions — Stroke | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Experimental): Simvastatin 40 mg daily for 3 months.
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40 mgrs daily for three months.

SUMMARY:
The purpose of this study is to determine whether simvastatin treatment started within the first 12 hours from stroke onset improves neurological and functional outcomes, evaluated at seventh day/discharge or at the third month.

Also, to demonstrate that simvastatin is safe and not associated with higher rates of hemorrhagic transformation in patients who receive thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years acute ischemic stroke (less than 12 hours from stroke onset).
* Stroke involving MCA-ACA-PCA.
* NIHSS score 4 to 22.
* Previous modified Rankin Scale score of 1 or 0.
* Patient or proxy informed consent.
* Patients not taking statins for the past six months.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Clinical or radiological evidence on admission of intracranial hemorrhage, hemorrhagic infarction or tumor.
* Seizures at the time of inclusion.
* Complete or substantial recovery prior to randomization.
* Patients with ipsilateral neurological deficit that may mask the evaluation of the current event.
* Liver disease (AST or ALT more than twice upper normality limit).
* Cardiogenic shock or relevant cardiac failure.
* Patients with more than five times upper normality limit of CPK.
* Myocardial infarction or any other thromboembolic event within the previous 30 days.
* Active infection by the time of inclusion.
* Documented hypersensibility to statins.
* Drug abuse.
* Expected short life-expectancy related to other systemic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is to determine whether simvastatin treatment started within the first 12 hours from stroke onset improves neurological and functional outcomes, evaluated at seventh day/discharge or at the third month. | Seventh day (or discharge) and third month

SECONDARY OUTCOMES:
The secondary outcome of this study is to demonstrate that simvastatin is safe and not associated with higher rates of hemorrhagic transformation in patients who receive thrombolysis. | 24 to 78 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joan Montaner, MD, PhD, Study Director — Hospital Vall Hebron Research Institute; Marc Ribó, MD, PhD, Principal Investigator — Hospital Vall Hebron. Stroke Unit; Carmen Jimenez, MD, Principal Investigator — Hospital Son Dureta. Stroke Unit.; Francesc Muñoz, MD, Principal Investigator — Hospital de Mollet; David Canovas, MD, Principal Investigator — Consorci Sanitari Parc Taulí Sabadell.; Jurek Krupinski, MD, Principal Investigator — Hospital Mutua de Terrassa. Neurology Department; Maite Martinez-Zabaleta, MD, Principal Investigator — Hospital de Donostia. Neurology Department; Francisco Javier De la Torre Laviana, MD, Principal Investigator — Hospital Virgen del Rocio. Stroke Unit.; Marimar Freijo, MD, Principal Investigator — Hospital de Basurto; Tomás Segura, MD, Principal Investigator — Hospital Universitario de Albacete; Juan Arenillas, MD, PhD, Principal Investigator — Hospital Universitario de Valladolid; Jose Manuel Flores, MD, Principal Investigator — Hospital de Ciudad Real; Francisco Alonso, MD, PhD, Principal Investigator — Hospital General de Vic; Jaime Masjuán Vallejo, MD, Principal Investigator — Hospital Universitario Ramón y Cajal. Stroke unit.; Francisco Rubio Borrego, MD, PhD, Principal Investigator — Hospital Universitario de Bellvitge. Stroke Unit.; Javier Tejada García, MD, Principal Investigator — Hospital de Leon; Aida Lago Martín, MD, PhD, Principal Investigator — Hospital Universitario la Fe. Stroke Unit.; Yolanda Bravo Anguiano, MD, Principal Investigator — Hospital General Yagüe; Xavier Ustrell Roig, MD, PhD, Principal Investigator — Hospital Universitario Joan XXIII; Francisco Purroy García, MD, PhD, Principal Investigator — Hospital Universitario Arnau de Vilanova de Lleida; Raquel Delgado Mederos, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (20):
- Spain (20):
  - Hospital General de Vic, Vic, Barcelona
  - Hospital Universitario de Albacete, Albacete
  - Hospital de Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital General Yagüe, Burgos
  - Hospital de Ciudad Real, Ciudad Real
  - Hospital de Donostia, Donostia / San Sebastian
  - Hospital de León, León
  - Hospital Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital de Mollet, Mollet del Vallès
  - Hospital Son Dureta, Palma de Mallorca
  - Consorci Sanitari Parc Tauli, Sabadell
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario Joan XXIII, Tarragona
  - Hospital Mutua de Terrassa, Terrassa
  - Hospital Universitario La Fe, Valencia
  - Hospital Universitario de Valladolid, Valladolid

REFERENCES:
- [Derived] Montaner J, Bustamante A, Garcia-Matas S, Martinez-Zabaleta M, Jimenez C, de la Torre J, Rubio FR, Segura T, Masjuan J, Canovas D, Freijo M, Delgado-Mederos R, Tejada J, Lago A, Bravo Y, Corbeto N, Giralt D, Vives-Pastor B, de Arce A, Moniche F, Delgado P, Ribo M; STARS Investigators. Combination of Thrombolysis and Statins in Acute Stroke Is Safe: Results of the STARS Randomized Trial (Stroke Treatment With Acute Reperfusion and Simvastatin). Stroke. 2016 Nov;47(11):2870-2873. doi: 10.1161/STROKEAHA.116.014600. Epub 2016 Oct 6. PMID 27758944